CLINICAL TRIAL: NCT03696732
Title: The Effect of Preoperative Anxiety on Phenylephrine Dosage During Cesarean Delivery Under Spinal Anesthesia, A Prospective Observational Study.
Brief Title: Anxiety and Phenylephrine Dosage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Associate Professor, Rabin Medical Center
Other Study IDs: 450-18
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Phenylephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing cesarean section: Women undergoing cesarean section under spinal anesthesia with prophylactic phenylephrine drip.
  Interventions: Other: Anxiety questionnaire; Other: VAS questionnaire

INTERVENTIONS:
Other: Anxiety questionnaire — Spielberger. State-Trait Inventory questionnaire
Other: VAS questionnaire — verbal numerical scale (VNS) anxiety score

SUMMARY:
Spinal anesthesia is considered gold standard anesthetic technique of choice for cesarean delivery (1). However its use is frequently associated with maternal hypotension, which occurs in up to 71% of cases, without prophylactic treatment(2) Spinal hypotension can lead to unpleasant maternal side effects such as nausea, vomiting and dizziness. In addition, adverse effects on the neonate occur because of reduced uteroplacental blood flow resulting in impaired fetal oxygenation and fetal acidosis. As such, current research recommends the prophylactic use of vasopressors for improved maternal and fetal outcomes(3).

The international consensus statement on the management of hypotension during cesarean delivery states, that a prophylactic phenylephrine infusion is superior to bolus administration and should be dose titrated according to blood pressure parameters (4). In according to the international guidelines, in our obstetric anesthesia unit, we use a standardized spinal anesthetic regime protocol with a standardized prophylactic phenylephrine infusion at a rate of 50 mcg/min, with the vasopressor dose titrated according to every minute blood pressure parameters.

Spinal anesthesia causes maternal hypotension, resulting from a blockade of sympathetic efferent neurons. Patients with higher baseline sympathetic activation have been known to have more marked hypotension after spinal anesthesia (5, 6) Anxiety causes generalized sympathetic activation (7). In a previous research the investigators showed that preoperative anxiety assessed by VAS had a significant effect on hypotension after spinal anesthesia (8).

Study objective:

In this study the investigators aim to evaluate the effect of anxiety on the cumulative phenylephrine dosage in women undergoing cesarean delivery under spinal anesthesia with prophylactic phenylephrine infusion. The primary hypothesis is that parturients who suffer from preoperative anxiety measured by a verbal numerical scale (VNS) anxiety score and Spielberger State-Trait Inventory questionnaire, will receive higher cumulative doses of phenylephrine (resulting from higher incidence of maternal hypotension).

DETAILED DESCRIPTION:
Methods:

This is a prospective, observational, single center study, which will be conducted at the Rabin Medical Center (Beilinson campus), Petach Tikva, Israel, a tertiary university hospital. This study Is a purely observational study, with no implication on the medical treatment provided.

Two hundred women aged 18 and above undergoing cesarean section delivery under spinal anesthesia will be enrolled after filling out an informed consent prior to surgery. Women will be requested to fill out an informed consent in the women's surgery waiting room on the day of surgery, when they aren't under any pain.

The parturients preoperative anxiety will be assessed in the women's waiting room, on the day of the surgery using two previously validated direct psychological measures of anxiety: verbal numerical scale (VNS) anxiety score (9, 10), and the Spielberger. State-Trait Inventory questionnaire (13).

Women will also be asked about nausea and vomiting during the surgery and in the post anesthesia care unit.

In according to standard departmental clinical practice, baseline blood pressure will be determined in the preoperative holding area by recording 3 times ≥ 3 minutes apart using an automated oscillometric blood pressure cuff on the arm with the patient supine with left uterine displacement, with the mean of the 3 values taken as a baseline systolic and diastolic blood pressure. Women will undergo spinal anesthesia and blood pressure will be measured evert minute during labor. Hypotension will be treated by titrating the phenylephrine infusion and by phenylephrine boluses, using a standardized algorithm according to departmental protocol. At the time of spinal injection, a phenylephrine infusion will be started at 50 mcg/min. The automated blood pressure cuff will be programmed to cycle each minute. When each new blood pressure result will appear, the phenylephrine infusion will be adjusted based on the systolic blood pressure by a standard algorithm.

Parturient's obstetric history, obstetric data and anesthetic data will be collected from each of the participant's medical file, in an anonymized way.

ELIGIBILITY:
Inclusion Criteria:

Healthy parturients undergoing cesarean delivery under spinal anesthesia in Beilinson Hospital.

Exclusion Criteria:

1. Women in active labor
2. Women with a twin pregnancy
3. Women with chronic hypertension or hypertension or preeclampsia.
4. Active medical or psychiatric disorders requiring regular medication.
5. Women who have any contraindication for spinal anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Two hundred healthy term parturients, over 18 years old, with healthy singleton pregnancy, undergoing cesarean delivery under spinal anesthesia in Beilinson Hospital, following obtaining written informed consents forums with the ability to comply with the study requirements will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Total cumulative phenylephrine dosage in women undergoing cesarean delivery under spinal anesthesia with prophylactic phenylephrine infusion. | During surgery -2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Reynolds F, Seed PT. Anaesthesia for Caesarean section and neonatal acid-base status: a meta-analysis. Anaesthesia. 2005 Jul;60(7):636-53. doi: 10.1111/j.1365-2044.2005.04223.x. PMID 15960713
- [Background] Higgins N, Fitzgerald PC, van Dyk D, Dyer RA, Rodriguez N, McCarthy RJ, Wong CA. The Effect of Prophylactic Phenylephrine and Ephedrine Infusions on Umbilical Artery Blood pH in Women With Preeclampsia Undergoing Cesarean Delivery With Spinal Anesthesia: A Randomized, Double-Blind Trial. Anesth Analg. 2018 Jun;126(6):1999-2006. doi: 10.1213/ANE.0000000000002524. PMID 28953494
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Hanss R, Bein B, Ledowski T, Lehmkuhl M, Ohnesorge H, Scherkl W, Steinfath M, Scholz J, Tonner PH. Heart rate variability predicts severe hypotension after spinal anesthesia for elective cesarean delivery. Anesthesiology. 2005 Jun;102(6):1086-93. doi: 10.1097/00000542-200506000-00005. PMID 15915018
- [Background] Hanss R, Ohnesorge H, Kaufmann M, Gaupp R, Ledowski T, Steinfath M, Scholz J, Bein B. Changes in heart rate variability may reflect sympatholysis during spinal anaesthesia. Acta Anaesthesiol Scand. 2007 Nov;51(10):1297-304. doi: 10.1111/j.1399-6576.2007.01455.x. PMID 17944631
- [Background] Roth WT, Doberenz S, Dietel A, Conrad A, Mueller A, Wollburg E, Meuret AE, Barr Taylor C, Kim S. Sympathetic activation in broadly defined generalized anxiety disorder. J Psychiatr Res. 2008 Feb;42(3):205-12. doi: 10.1016/j.jpsychires.2006.12.003. Epub 2007 Jan 23. PMID 17250853
- [Background] Orbach-Zinger S, Ginosar Y, Elliston J, Fadon C, Abu-Lil M, Raz A, Goshen-Gottstein Y, Eidelman LA. Influence of preoperative anxiety on hypotension after spinal anaesthesia in women undergoing Caesarean delivery. Br J Anaesth. 2012 Dec;109(6):943-9. doi: 10.1093/bja/aes313. Epub 2012 Sep 10. PMID 22964265
- [Background] Vogelsang J. The Visual Analog Scale: an accurate and sensitive method for self-reporting preoperative anxiety. J Post Anesth Nurs. 1988 Aug;3(4):235-9. No abstract available. PMID 2457102
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461